CLINICAL TRIAL: NCT05711147
Title: One-time Abutment Placement Versus 4 Times Abutment Removal on Interproximal Bone Levels and Peri-implant Soft Tissues: a Prospective Randomized Clinical Trial
Brief Title: One-time Abutment Placement Versus 4 Times Abutment Removal Around Dental Implants
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Camlog Oral Reconstruction Foundation (Other)
Responsible Party: Principal Investigator, Ana Molina Villar, Assistant Professor, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17/291-R_X
Record Dates: First submitted 2023-01-24; First posted 2023-02-02 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Dental Implant; Prosthetic Abutment

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Definitive abutment (Experimental): Definitive prosthetic abutment placed at the moment of implant placement
  Interventions: Procedure: Placement of definitive abutment
- Healing abutment (Active Comparator): Conventional healing abutment placed at the moment of implant placement and removed 4 times during prosthesis making
  Interventions: Procedure: Abutment removal

INTERVENTIONS:
Procedure: Abutment removal — 4 times healing abutment removal during prosthesis making (impressions, metal try-in, ceramic try-in, prosthesis loading)
  Arms: Healing abutment
Procedure: Placement of definitive abutment — Placement of the final prosthetic abutment at the moment of implantation
  Arms: Definitive abutment

SUMMARY:
Introduction: the repeated connection and disconnection of healing abutments during dental implants´ osseointegration has been associated with significant increased peri-implant bone loss, when compared with placing the final prosthetic abutment during implant placement surgery and non-removing it ever again. Previous data from animal studies suggests that the higher the number of removals of the healing abutments, the greater the bone resorption around implants, however the evidence in humans is scarce and heterogeneous. Furthermore, this greater bone resorption has been claimed to be associated to the inflammatory status of the peri-implant soft tissues, which would be greater as a consequence of the repeated disruption of the soft-tissues attachment to the prosthetic abutment, and the hypothetical microbial contamination of the implant-abutment interphase, induced by the repeated manipulation of the prosthetic components.

Objective: to evaluate the changes in peri-implant crestal bone levels between two prosthetic protocols, the control being the conventional protocol where healing abutments are placed during surgery and removed four times before the delivery of the final abutment and prostheses, and the test protocol where definitive abutments are placed immediately after implant placement and are not removed ever again.

Material and methods: 80 platform switched implants will be placed in the posterior maxilla or mandible of 40 partial edentulous patients. Immediately after implant placement, patients will be randomized to receive the definitive abutment at the moment of implant placement (one abutment-one time protocol), or 12 weeks later, after removing the healing abutment four times during the confection of the final prostheses, following the conventional protocol for implant supported restorations. The day of prostheses delivery, a mucosal biopsy from the implant surrounding tissues will be taken for histomorphometric and immunohistochemical analyses of the inflammatory response of the peri-implant soft tissues. Radiographic assessment of vertical bone level changes (primary outcome), clinical status of peri-implant tissues, changes in soft tissues margin, patient related outcomes and adverse events will be assessed at 6, 12, 24 and 36 months after loading.

ELIGIBILITY:
Inclusion Criteria:

* At least two adjacent missing teeth in the posterior maxilla or mandible (positions 4 to 7)
* Willing to receive implant supported fixed partial dentures
* There must be a natural tooth mesial to the most proximal implant site, however free end situations will be allowed for the distal implants
* Healed sites (minimum 12 weeks post-extraction)
* In the case of prior bone augmentation, a minimum of 6 months of healing is required
* Simultaneous bone augmentation will be allowed only for close sinus lifting

Exclusion Criteria:

Systemic exclusion criteria:

* Medical conditions requiring prolonged use of steroids and/or medications that can interfere with bone metabolism
* History of leukocyte dysfunction and deficiencies
* History of neoplastic disease requiring the use of radiation or chemotherapy
* History of renal failure
* Metabolic disorders such as osteoporosis
* History of uncontrolled endocrine disorders
* Physical handicaps that would interfere with the ability to perform adequate oral hygiene
* Alcoholism or drug abuse
* History of immunodeficiency syndromes
* Smokers of >10 cigarettes per day, cigar equivalents or tobacco chewers
* Any other condition or circumstance that, in the opinion of the investigator, would prevent completion of the study participation or interfere with the analysis of the study results, such as history of non-compliance or unreliability

Local exclusion criteria:

* Any kind of bone augmentation performed on the implant site, with a healing period of <6 months
* Local inflammation (including untreated periodontitis)
* Mucosal diseases such as erosive liquen planus
* Less than 2mm of keratinized mucosa in the intended implant sites
* History of local irradiation therapy
* Presence of osseous lesions
* History of implant failure
* Post-extraction sites with <12 weeks of healing
* Severe bruxism or clenching habits
* Persistent intraoral infection

Exclusion criteria at surgery: in any of the following circumstances, the patient will not be randomized and will be excluded from the analysis

* Lack of primary stability at surgery
* Need for crestal augmentation procedures during implant surgery
* Inability to place the implants according to the prosthetic requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Changes in interproximal bone levels | Implantation, prosthesis loading, 6 months, 12 months, 24 months, 36 months
  Changes at the mesial and distal crestal bone levels measured in periapical digital radiographs at the mesial and distal implant aspects

SECONDARY OUTCOMES:
Mobility | Prosthesis loading, 6 months, 12 months, 24 months, 36 months
  Implant and/or prostheses mobility
Keratinized peri-implant mucosa | Prosthesis loading, 6 months, 12 months, 24 months, 36 months
  Presence or absence of keratinized peri-implant mucosa in the mid-buccal and mid-lingual aspects
Modified plaque index | Prosthesis loading, 6 months, 12 months, 24 months, 36 months
  Modified plaque index (Mombelli et al. 1987) at six sites per implant
Sulcus bleeding index | Prosthesis loading, 6 months, 12 months, 24 months, 36 months
  Sulcus bleeding index (Mombelli et al. 1987) at six sites per implant
Probing depth | Prosthesis loading, 6 months, 12 months, 24 months, 36 months
  Probing depth (Mombelli et al. 1987) at six sites per implant
Clinical crown length of the adjacent tooth | Prosthesis loading, 6 months, 12 months, 24 months, 36 months
  CLT: distance in mm from the highest line of gingival/mucosal curvature of the crown to the occlusal aspect of the tooth
Clinical crown length of the implant supported crown | Prosthesis loading, 6 months, 12 months, 24 months, 36 months
  CLI: distance in mm from the highest line of mucosal curvature of the crown to the occlusal aspect of the implant prostheses
Papilla index | Prosthesis loading, 6 months, 12 months, 24 months, 36 months
  IP: distance in mm from the top of the mesial and distal papillae of each implant to the most coronal portion of the contact point or the occlusal surface (Grunder 2000)
Patient-reported outcomes | Prosthesis loading, 6 months, 12 months, 24 months, 36 months
  5-items questionnaire (comfort, appearance, masticatory function, taste and overall satisfaction) rated according to the following scale: very unsatisfied, unsatisfied, fair, satisfied, and very satisfied
Adverse events | Prosthesis loading, 6 months, 12 months, 24 months, 36 months
  Occurrence and nature of adverse events, either "implant or prostheses associated" (device related adverse events and other tissue complications), or "non-implant associated" (death, serious illness or any condition requiring hospitalization for more than 1 day).
Hystomorphometric analysis of soft tissue biopsy samples | Prosthesis loading
  Total areas of the sample, the epithelium, the connective tissue, the inflammatory infiltrate and cell density in an interest area into the inflammatory infiltrate
Immunohistochemical analysis of the histologic sections | Prosthesis loading
  Nature and extension of the inflammatory infiltrate in the connective tissue: high positive (HP), positive (P), low positive (LP) or negative (N) staining

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Sanz, Prof. Dr., Principal Investigator — University Complutense of Madrid
Locations (1):
- Dental School, University Complutense of Madrid, Madrid, Spain